CLINICAL TRIAL: NCT00000960
Title: A Phase III Randomized Placebo-Controlled Trial to Evaluate the Efficacy, Safety and Tolerance of Oral Zidovudine (AZT) in Pregnant HIV Infected Women and Their Infants
Brief Title: The Safety and Effectiveness of Zidovudine in HIV-Infected Pregnant Women and Their Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Glaxo Wellcome (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 076; 11050 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Pregnancy
Keywords: Pregnancy; Pregnancy Complications, Infectious; Prenatal Exposure Delayed Effects; Administration, Oral; AIDS-Related Complex; Zidovudine
MeSH Terms: conditions — HIV Infections; Pregnancy Complications, Infectious; Prenatal Exposure Delayed Effects; AIDS-Related Complex | interventions — Zidovudine

INTERVENTIONS:
Drug: Zidovudine

SUMMARY:
To determine whether the rate of HIV transmission from mother to infant can be reduced by continuous oral zidovudine (AZT) treatment to HIV infected pregnant women, intravenous AZT during childbirth, and oral AZT treatment of the newborn infant from birth to six weeks of age. The study is also designed to evaluate the safety of AZT for both the pregnant woman and the newborn infant.

No method exists to prevent transmission of HIV from an infected mother to her newborn infant. Giving an antiviral agent (such as AZT) to the mother and to the newborn could in theory decrease the risk of infection to the newborn by reducing the exposure of the fetus to maternal virus, or by preventive treatment of the fetus before exposure.

DETAILED DESCRIPTION:
No method exists to prevent transmission of HIV from an infected mother to her newborn infant. Giving an antiviral agent (such as AZT) to the mother and to the newborn could in theory decrease the risk of infection to the newborn by reducing the exposure of the fetus to maternal virus, or by preventive treatment of the fetus before exposure.

Patients are enrolled during their pregnancy, between 14 and 34 weeks of gestation. They are chosen by random selection to receive AZT or placebo. Treatment continues until labor at which time they begin to receive continuous intravenous study drug. Study drug treatment is discontinued after the umbilical cord is clamped. AZT is then offered all women as per labeled indications for 6 weeks postpartum, while appropriate medical followup is being arranged. Mothers who develop an AIDS defining illness or whose CD4+ cell counts decrease to less than 200 cells/mm3 during pregnancy are offered open-label drug at that time. The mother is followed by her primary obstetrician at an AIDS Clinical Trials Unit (ACTU) or subunit facility. The mother may deliver at the ACTU or a non-ACTU site. Treatment of the infant is started in the newborn nursery and continues on an outpatient basis. Infants receive the same study treatment as the mother for 6 weeks, and are monitored to week 78.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed for infants:

* Treatment for signs of drug withdrawal (e.g., phenobarbital, chlorpromazine, tincture of opium, paregoric, or Valium).
* Treatment for nonserious conditions (e.g., syphilis treatment, hepatitis B vaccine).
* All essential supportive treatment for conditions that are nonlife threatening as deemed by the on-site pediatrician.
* Acetaminophen.
* Standard immunizations.
* Allowed for women:
* All medications/treatments as required for normal OB care of HIV+ women, except as noted under exclusions.
* Pneumocystis prophylaxis as indicated.
* Topical steroids. Parenteral and oral steroids for 6 or fewer days.

Concurrent Treatment:

Allowed for pregnant woman:

Blood transfusion for anemia (hemoglobin less than 7 g/dl).

Allowed for infant:

- Blood transfusions for anemia except if attributed to study drug.

-

Patients must:

* Have HIV infection.
* Intend to carry pregnancy to term.
* Be willing to be followed by a participating ACTG center for duration of the study.
* Be able to provide informed consent (if available, father of the fetus must also provide informed consent).
* Infants may enroll simultaneously in other pediatric protocols after completing the initial 6 weeks of study treatment.
* Inclusion age for women is 13 years old or more or IRB local age of consent.
* Inclusion age for infants is 0 to 20 months.

Exclusion Criteria

Co-existing Condition:

Infants with the following conditions or symptoms are excluded:

* Requiring treatment for hyperbilirubinemia (except phototherapy).

Concurrent Medication:

Excluded:

* Infants:
* Antiretroviral drugs or vaccines.
* Excluded during current pregnancy:
* Zidovudine (AZT).
* Other antiretroviral agents (e.g., rCD4, CD4-IgG, d4T, didanosine (ddI), dideoxycytidine (ddC)), passive immunotherapy (e.g., HIVIG), anti-HIV vaccines, cytolytic chemotherapeutic agents.
* Corticosteroids for equal to or more than 7 days.

Patients with the following are excluded:

* Evidence of preexisting fetal anomalies that may (1) result in a high probability that the fetus/infant will not survive to the end of the study period (e.g., anencephaly, renal agenesis, or Potter's syndrome); or (2) increase the fetal tissue concentration of zidovudine (AZT) or its metabolites to a toxic level (e.g., neural tube or ventral wall defects).
* Baseline sonogram completed within 28 days prior to randomization that demonstrates 2nd trimester findings of anencephaly or oligohydramnios, or 3rd trimester findings of unexplained polyhydramnios, fetal hydrops, ascites or other evidence of preexisting in-utero anemia.
* History of intolerance to AZT dose of 500 or less mg/day prior to this pregnancy that resulted in discontinuation of treatment for more than 4 weeks.
* Recipient of AZT during current pregnancy for any indication or meet criteria for AZT as defined by this protocol (CD4+ cell counts less than 200 cells/mm3 or AIDS).
* Infants not having parent/guardian available to give informed consent if necessary.

Prior Treatment:

Excluded during current pregnancy:

* Radiation therapy.

Ages: 1 Day to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1496
Dates: Study Completion 1994-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E Connor, Study Chair; R Sperling, Study Chair
Locations (62):
- United States (58):
  - Univ of Alabama at Birmingham Schl of Med / Pediatrics, Birmingham, Alabama
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - UCSD Med Ctr / Pediatrics / Clinical Sciences, La Jolla, California
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - UCLA Med Ctr / Pediatric, Los Angeles, California
  - Harbor - UCLA Med Ctr / UCLA School of Medicine, Los Angeles, California
  - San Francisco Gen Hosp, San Francisco, California
  - Children's Hosp of Denver, Denver, Colorado
  - Univ of Connecticut / Farmington, Farmington, Connecticut
  - Univ of Connecticut Health Ctr, Farmington, Connecticut
  - Howard Univ Hosp, Washington D.C., District of Columbia
  - Univ of Miami (Pediatric), Miami, Florida
  - Northwestern Univ Med School, Chicago, Illinois
  - Cook County Hosp, Chicago, Illinois
  - Univ of Illinois College of Medicine / Pediatrics, Chicago, Illinois
  - Chicago Children's Memorial Hosp, Chicago, Illinois
  - Univ of Chicago Children's Hosp, Chicago, Illinois
  - Tulane Univ / Charity Hosp of New Orleans, New Orleans, Louisiana
  - Univ of Maryland at Baltimore / Univ Med Ctr, Baltimore, Maryland
  - Johns Hopkins Hosp - Pediatric, Baltimore, Maryland
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Children's Hosp of Boston, Boston, Massachusetts
  - Boston City Hosp / Pediatrics, Boston, Massachusetts
  - Beth Israel Deaconess Med Ctr, Boston, Massachusetts
  - Baystate Med Ctr of Springfield, Springfield, Massachusetts
  - Univ of Massachusetts Med Ctr, Worcester, Massachusetts
  - Children's Hosp of Michigan, Detroit, Michigan
  - UMDNJ - New Jersy Med School, Newark, New Jersey
  - Univ of Medicine & Dentistry of New Jersey / Univ Hosp, Newark, New Jersey
  - Children's Hosp of New Jersey / UMDNJ - New Jersey Med Schl, Newark, New Jersey
  - Children's Hosp at Albany Med Ctr, Albany, New York
  - SUNY - Brooklyn, Brooklyn, New York
  - SUNY / Health Sciences Ctr at Brooklyn / Pediatrics, Brooklyn, New York
  - Beth Israel Med Ctr / Pediatrics, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Cornell Univ Med College, New York, New York
  - Mount Sinai Med Ctr / Pediatrics, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - State Univ of New York at Stony Brook, Stony Brook, New York
  - SUNY Health Sciences Ctr at Syracuse / Pediatrics, Syracuse, New York
  - Bronx Lebanon Hosp Ctr, The Bronx, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Westchester Hosp, Valhalla, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Carolinas Med Ctr, Charlotte, North Carolina
  - Duke Univ Med Ctr, Durham, North Carolina
  - Univ of Cincinnati, Cincinnati, Ohio
  - Children's Hosp of Philadelphia, Philadelphia, Pennsylvania
  - Hosp of the Univ of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson Univ Hosp, Philadelphia, Pennsylvania
  - Rhode Island Hosp / Brown Univ, Providence, Rhode Island
  - Med Univ of South Carolina, Charleston, South Carolina
  - Saint Jude Children's Research Hosp of Memphis, Memphis, Tennessee
  - Children's Med Ctr of Dallas, Dallas, Texas
  - Lyndon Baines Johnson Gen Hosp, Houston, Texas
  - Texas Children's Hosp / Baylor Univ, Houston, Texas
  - Children's Hosp of Seattle, Seattle, Washington
- Puerto Rico (4):
  - Ramon Ruiz Arnau Univ Hosp / Pediatrics, Bayamón
  - Univ of Puerto Rico / Univ Children's Hosp AIDS, San Juan
  - UPR Children's Hosp / UPR School of Medicine, San Juan
  - San Juan City Hosp, San Juan

REFERENCES:
- [Background] Sperling RS, Shapiro DE, Coombs RW, Todd JA, Herman SA, McSherry GD, O'Sullivan MJ, Van Dyke RB, Jimenez E, Rouzioux C, Flynn PM, Sullivan JL. Maternal viral load, zidovudine treatment, and the risk of transmission of human immunodeficiency virus type 1 from mother to infant. Pediatric AIDS Clinical Trials Group Protocol 076 Study Group. N Engl J Med. 1996 Nov 28;335(22):1621-9. doi: 10.1056/NEJM199611283352201. PMID 8965861
- [Background] Connor EM, Sperling RS, Gelber R, Kiselev P, Scott G, O'Sullivan MJ, VanDyke R, Bey M, Shearer W, Jacobson RL, et al. Reduction of maternal-infant transmission of human immunodeficiency virus type 1 with zidovudine treatment. Pediatric AIDS Clinical Trials Group Protocol 076 Study Group. N Engl J Med. 1994 Nov 3;331(18):1173-80. doi: 10.1056/NEJM199411033311801. PMID 7935654
- [Background] Sperling RS, Shapiro DE, McSherry GD, Britto P, Cunningham BE, Culnane M, Coombs RW, Scott G, Van Dyke RB, Shearer WT, Jimenez E, Diaz C, Harrison DD, Delfraissy JF. Safety of the maternal-infant zidovudine regimen utilized in the Pediatric AIDS Clinical Trial Group 076 Study. AIDS. 1998 Oct 1;12(14):1805-13. doi: 10.1097/00002030-199814000-00012. PMID 9792381
- [Background] Wiznia AA, Crane M, Lambert G, Sansary J, Harris A, Solomon L. Zidovudine use to reduce perinatal HIV type 1 transmission in an urban medical center. JAMA. 1996 May 15;275(19):1504-6. PMID 8622226
- [Background] Rouzioux C. Prevention of maternal HIV transmission. Practical guidelines. Drugs. 1995;49 Suppl 1:17-24; discussion 38-40. doi: 10.2165/00003495-199500491-00006. PMID 7614898
- [Background] Dickover RE, Garratty EM, Herman SA, Sim MS, Plaeger S, Boyer PJ, Keller M, Deveikis A, Stiehm ER, Bryson YJ. Identification of levels of maternal HIV-1 RNA associated with risk of perinatal transmission. Effect of maternal zidovudine treatment on viral load. JAMA. 1996 Feb 28;275(8):599-605. PMID 8594240
- [Background] Culnane M, Fowler M, Lee SS, McSherry G, Brady M, O'Donnell K, Mofenson L, Gortmaker SL, Shapiro DE, Scott G, Jimenez E, Moore EC, Diaz C, Flynn PM, Cunningham B, Oleske J. Lack of long-term effects of in utero exposure to zidovudine among uninfected children born to HIV-infected women. Pediatric AIDS Clinical Trials Group Protocol 219/076 Teams. JAMA. 1999 Jan 13;281(2):151-7. doi: 10.1001/jama.281.2.151. PMID 9917118
- [Background] Shearer WT, Quinn TC, LaRussa P, Lew JF, Mofenson L, Almy S, Rich K, Handelsman E, Diaz C, Pagano M, Smeriglio V, Kalish LA. Viral load and disease progression in infants infected with human immunodeficiency virus type 1. Women and Infants Transmission Study Group. N Engl J Med. 1997 May 8;336(19):1337-42. doi: 10.1056/NEJM199705083361901. PMID 9134873
- [Background] Frenkel LM, Cowles MK, Shapiro DE, Melvin AJ, Watts DH, McLellan C, Mohan K, Murante B, Burchett S, Bryson YJ, O'Sullivan MJ, Mitchell C, Landers D. Analysis of the maternal components of the AIDS clinical trial group 076 zidovudine regimen in the prevention of mother-to-infant transmission of human immunodeficiency virus type 1. J Infect Dis. 1997 Apr;175(4):971-4. doi: 10.1086/514003. PMID 9086162
- [Background] Newell ML, Gray G, Bryson YJ. Prevention of mother-to-child transmission of HIV-1 infection. AIDS. 1997;11 Suppl A:S165-72. No abstract available. PMID 9451981
- [Result] Edathodu J, Halim MM, Dahham MB, Alrajhi AA. Mother-to-child transmission of HIV: experience at a referral hospital in Saudi Arabia. Ann Saudi Med. 2010 Jan-Feb;30(1):15-7. doi: 10.4103/0256-4947.59367. PMID 20103953